CLINICAL TRIAL: NCT02706314
Title: Pilot Observation of the Impact of Human Blood Serum From Critically Ill Patients With or Without Critical-illness-polyneuropathy on Intramural Neuronal Networks of Human Colon Samples
Brief Title: Impact of Human Blood Serum From Critically Ill Patients on Human Colon Neuronal Networks.
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dr. Johannes Ehler, MD, Dr. med. Johannes Ehler, University of Rostock
Other Study IDs: A 2016-0016
Record Dates: First submitted 2016-02-23; First posted 2016-03-11 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Critical Illness; Multiple Organ Failure; Polyneuropathy; Myopathy
MeSH Terms: conditions — Critical Illness; Multiple Organ Failure; Polyneuropathies; Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum probes will be stored at -80°C.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Critically ill patients with CIP: Critically ill patients with a Sequential Organ Failure Assessment (SOFA)-Score >7 with CIP
- Critically ill patients without CIP: Critically ill patients with a Sequential Organ Failure Assessment (SOFA)-Score >7 without CIP
- Healthy volunteers: Healthy volunteers with neither critical illness nor CIP

SUMMARY:
Critical illness in the ICU setting has high medical and socioeconomic importance. Critically ill patients frequently develop severe neurologic impairment during their course of disease, typically presenting as critical-illness-polyneuropathy (CIP), which is associated with an increased mortality rate. To date neither strategies are available to predict nor to specifically treat CIP.

Diagnostic tests to determine CIP during the course of critical illness are available through nerve conduction studies. Further research is needed to find diagnostic tools to identify patients who are on high risk to develop CIP, which could encourage the evolution of new therapeutic strategies for CIP patients.

The aims of the study are:

1. An early detection of changes in intramural neuronal networks of human colon samples induced by human blood serum from critically ill patients in order to predict the development of CIP
2. The comparison of different diagnostic tests to diagnose and monitor CIP during the course of critical illness (neurologic examination versus nerve conduction study versus neuromyosonography)

DETAILED DESCRIPTION:
All patients with critical illness and fulfilling the inclusion criteria should be screened for the study on two surgical ICUs at the university hospital of Rostock, Germany.

The inclusion of patients will be started if written informed consent was obtained from all participants or their representatives (if direct consent could not be obtained).

The aim of the study is a prediction or an earlier detection of CIP in critically ill patients before nerve conduction studies are able to diagnose CIP. We hypothesize that upregulated circulating neurotoxic factors in human serum of critically ill patients cause neuronal damage and play an important role in the pathogenesis of CIP. Time from upregulation of neurotoxic factors to the clinical appearance of neuronal damage (CIP) is unknown.

An experimental part of the study aims at establishing enteric neuronal networks as functional bioassays for the qualitative detection of neurotoxic humoral factors. Human colon samples will be exposed to the serum of critically ill patients with and without CIP in an organ bath (100% serum) under standardized physiologic conditions. Alterations to neuronal functions (contractions, spontaneous activity) will be studied between serum from patients with CIP, without CIP and serum probes from healthy volunteers (without critical illness).

In a clinical part of the study critically ill patients with and without CIP (detected by nerve conduction studies as the gold standard for the diagnosis of CIP) will be examined by neurologic examination, nerve conduction study and neuromyosonography of peripheral nerves. The incidence, the extent and the time from the beginning of critical illness to the clinical appearance of nerval alterations will be compared between the 3 diagnostic tests.

From all patients basic demographic data, illness severity scores (APACHE-II, SOFA) laboratory results, pre-morbidity data and clinical outcome for the study cohort will be recorded. At day 3 and 10 patients will be examined by neurologic examination, nerve conduction study, neuromyosonography and laboratory tests (inflammation, coagulation, organ function, blood parameters including TNF-alpha, IL-6, S100b, oxidative stress markers, neurofilaments, C-type natriuretic peptide).

ELIGIBILITY:
Inclusion Criteria:

* Patients with critical illness, defined as a SOFA-Score ≥ 8 on 3 consecutive days within the first 5 days of ICU stay
* Informed consent by patient or legal proxy

Exclusion Criteria:

* Diagnosis of pre-existing neuromuscular diseases other than CIP
* High-dose glucocorticosteroid therapy (> 300 mg Hydrocortisone/die)
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with critical illness and fulfilling the inclusion criteria should be screened for the study on two surgical ICUs at the university hospital of Rostock, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-03; Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Changes in the frequency and the amplitude of spontaneous contractions of colonic smooth muscle preparations induced by incubation with serum from critically ill patients with CIP, without CIP and healthy controls | Baseline and 3 Hours
  The parameters will be measured in colonic smooth muscle preparations before and after three hours of incubation with serum from healthy controls as well as critically ill patients with or without CIP. The observed changes in the respective parameter over the three-hour period will be estimated in each tested preparation as measured by absolute values of frequency (contractions per minute) and force (millinewton).
Changes in the amplitude, the integrated force and the time to first and last peak of contractions evoked by electric field stimulation in colonic smooth muscle preparations incubated with the above mentioned sera | Baseline and 3 Hours
  Applying the same time protocol as described above for point 1, except for the use of electric field stimulation as an exogenous trigger of contractions, changes in the respective parameter over the three-hour period will be estimated in each tested preparation as measured by absolute values of force (millinewton), integrated force (millinewton*second) and time (seconds).

SECONDARY OUTCOMES:
Incidence of CIP assessed by standardized nerve conduction study | Day 10
  CIP defined as a reduction in the amplitude of compound muscle action potentials and sensory nerve action potentials
Incidence of CIP assessed by standardized neurological examination | Day 10
  CIP defined as decreased or absent tendon reflexes and/or muscular paresis
Incidence of peripheral nerve abnormalities assessed by neuromyosonography | Day 10
  Defined as increased nerve cross sectional areas in mm²
Incidence of abnormalities of muscle echogenicity assesed by neuromyosonography | Day 10
  Abnormal muscle echogenicity defined as mild, moderate or massive increased echogenicity in comparison to bone echogenicity
Time of respirator-therapy | Day 100
Length of ICU stay | Day 100
The number of participants with death | Day 100

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit PIT 1 and 2, University hospital Rostock, Rostock, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klawitter F, Laukien F, Fischer DC, Rahn A, Porath K, Danckert L, Bajorat R, Walter U, Patejdl R, Ehler J. Longitudinal Assessment of Blood-Based Inflammatory, Neuromuscular, and Neurovascular Biomarker Profiles in Intensive Care Unit-Acquired Weakness: A Prospective Single-Center Cohort Study. Neurocrit Care. 2025 Feb;42(1):118-130. doi: 10.1007/s12028-024-02050-x. Epub 2024 Jul 9. PMID 38982001